CLINICAL TRIAL: NCT03374956
Title: Individualized Pharmacological Approach to Obesity Management: A Randomized Clinical Trial
Brief Title: Individualized Obesity Pharmacotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Andres J. Acosta, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-003449
Record Dates: First submitted 2017-11-09; First posted 2017-12-15 (Actual); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Obesity
Keywords: Pharmacological; Obesity Management; Individualized
MeSH Terms: conditions — Obesity | interventions — Qsymia; Liraglutide; Naltrexone; Bupropion; bupropion hydrochloride, naltrexone hydrochoride drug combination; Phentermine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Phenotype-guided pharmacotherapy, which includes Phentermine-Topiramate, Liraglutide, Naltrexone/bupropion or Phentermine plus Exercise
  Interventions: Drug: Phentermine-Topiramate; Drug: Liraglutide; Drug: Naltrexone/bupropion
- Control Group (Active Comparator): Randomly assigned pharmacotherapy, which includes Phentermine-Topiramate, Liraglutide, Naltrexone/bupropion or Phentermine
  Interventions: Drug: Phentermine-Topiramate; Drug: Liraglutide; Drug: Naltrexone/bupropion; Drug: Phentermine

INTERVENTIONS:
Drug: Phentermine-Topiramate — Extended Release at dose of 7.5/46 mg oral daily
  Other Names: Qsymia
Drug: Liraglutide — dose of 3 mg subcutaneous daily
  Other Names: Saxenda
Drug: Naltrexone/bupropion — Oral naltrexone extended-release/bupropion extended-release at dose of 32/360 mg oral daily (divided in 2 tables in morning and 2 tablets in evening)
  Other Names: Contrave
Drug: Phentermine — 15-37.5 mg oral daily
  Other Names: Adipex-P; Lomaira
  Arms: Control Group

SUMMARY:
The researchers are trying to identify the specific characteristics (phenotypes) that may be useful to help select the right medication for weight loss.

DETAILED DESCRIPTION:
All participants will be phenotype and participants will randomized to randomly assigned medications vs phenotype guided medications for obesity. All participants will receive a standard intense lifestyle intervention.All participants will be seen at 4 and 12 weeks. At the 12-week visit, participants will be unblinded to their "obesity-related phenotype" and they could contact their physician to continue a FDA-approved medication as part of clinical care. Study team will prospectively follow the patients' weight, waist circumference and use of obesity medications every 3 months for 1 year.

ELIGIBILITY:
Inclusion criteria:

* Adults with obesity (BMI >30 Kg/m2); these will be otherwise healthy individuals with no unstable psychiatric disease and controlled comorbidities or other diseases.
* Gender: Men or women. Women of childbearing potential will have negative pregnancy tests within 48 hours of enrollment and before each radiation exposure.

Exclusion criteria

* Abdominal bariatric surgery
* Positive history of chronic gastrointestinal diseases, or systemic disease that could affect gastrointestinal motility, or use of medications that may alter gastrointestinal motility, appetite or absorption, e.g., orlistat, within the last 6 months.
* Significant untreated psychiatric dysfunction based upon screening with the Hospital Anxiety and Depression Inventory (HAD), and the Questionnaire on Eating and Weight Patterns (binge eating disorders and bulimia). If such a dysfunction is identified by an anxiety or depression score >11 or difficulties with substance or eating disorders, the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up.
* Hypersensitivity to any of the study medications.
* No contraindications to all FDA-approved medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres J Acosta, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Acosta A, Camilleri M, Abu Dayyeh B, Calderon G, Gonzalez D, McRae A, Rossini W, Singh S, Burton D, Clark MM. Selection of Antiobesity Medications Based on Phenotypes Enhances Weight Loss: A Pragmatic Trial in an Obesity Clinic. Obesity (Silver Spring). 2021 Apr;29(4):662-671. doi: 10.1002/oby.23120. PMID 33759389
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 93 | 100
Completed | 93 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 93 | 100 | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 93 | 100 | 193
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (16) | 39 (14) | 39 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 78 | 143
  Male | 28 | 22 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 88 | 87 | 175
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 10 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 93 | 100 | 193

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Body Weight
Description: Percent change in body weight
Time Frame: baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 93 | 100
percent change | -7.7 [-11 to -4.7] | -6.5 [-11 to -2.3]

2. Secondary Outcome: Percentage of Responders
Description: Percentage of participants who loss 5% or more of total body weight
Time Frame: baseline to 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 93 | 100
percentage of participants | 81 | 80

3. Secondary Outcome: Percentage of Responders
Description: Percentage of participants with at least 10% total body weight loss
Time Frame: baseline to 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 93 | 100
percentage of participants | 44 | 40

ADVERSE EVENTS:
Time Frame: Baseline to 12 months
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/100
Other Adverse Events (participants affected / at risk) | 23/93 | 25/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=93) | Control Group (N=100)
During study (Gastrointestinal disorders) | 23 (23) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT03374956/Prot_SAP_001.pdf